CLINICAL TRIAL: NCT07230977
Title: A Phase I, Two-Part, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activities of GenSci139 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: GenSci139 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GenSci139-101
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part1 dose escalation (Experimental): dose escalation cohorts of GenSci139 in sequential ascending order
  Interventions: Drug: GenSci139
- Part 1 backfill (Experimental): backfill study at dose levels proved safety and efficacy during dose escalation
  Interventions: Drug: GenSci139
- Part 2 dose expansion (Experimental): Dose expansion at RDE dose levels with selected advanced cancers.
  Interventions: Drug: GenSci139

INTERVENTIONS:
Drug: GenSci139 — GenSci139 is a bispecific antibody drug conjugate targeting EGFR and HER2.

SUMMARY:
This is a phase I, two-part, multicenter, first-in-human study. The Part 1 study will assess the safety, tolerability, preliminary anti-tumor activities, PK profile, immunogenicity and biomarker of GenSci139 in participants with locally advanced or metastatic solid tumors, as well as identity MTD (if any) and RDE. The Part 2 study is to further evaluate the preliminary anti-tumor activities, safety, PK profile, immunogenicity and biomarker of GenSci139 at RDE dose levels with selected advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Has the ability to understand and the willingness to sign a written informed consent document (prior to the initiation dose of GenSci139 and any study procedures).
* Is willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other specified study procedures.
* Adult participants (≥18 years of age or acceptable age according to local regulations, whichever is older) at the time of voluntarily signing informed consent.
* Is able to provide tumor tissues. Fresh biopsy specimens or archival tumor tissue samples obtained after last treatment are strongly preferred, and if not available, providing other archival tumor tissue specimens or not may be enrolled after discussion with sponsor.
* Has at least one measurable lesion by RECIST v1.1.
* Has an eastern cancer collaboration group (ECOG) status of 0 or 1.
* Left ventricular ejection fraction (LVEF) ≥50%.
* Has a life expectancy of ≥ 3 months.
* Has adequate hematologic and organ function prior to initiation dose of GenSci139.
* Women of childbearing potential (WOCBP) must be willing to use adequate contraception while receiving GenSci139, and within 6 months after the last dose of GenSci139 and have a negative serum human chorionic gonadotropin (HCG) test.
* Nonsterile males must be willing to use adequate contraception for the duration of receiving GenSci139 and within 6 months after the last dose of GenSci139.
* Has histologically or cytologically confirmed locally advanced or metastatic UC, HNSCC, TNBC, NSCLC, BTC, ESCC, GC, CRC, OC, NPC, PDAC etc. and have progressed following standard therapy, or for whom, in the opinion of the investigator, no available and effective standard therapy exists.

Key Exclusion Criteria:

* Any active malignancy within 3 years before initiation dose of GenSci139 except for the cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, non-muscle invasive bladder cancer (NMIBC), carcinoma in situ of the cervix or breast).
* Has diagnosed as primary central nervous system (CNS) tumor.
* Has CNS metastases, unless asymptomatic, neurologically stable and not requiring steroids treatment for at least 4 weeks prior to initiation dose of GenSci139.
* Has a history of leptomeningeal disease or spinal cord compression.
* Has stroke or transient ischemic attack within 6 months prior to initiation dose of GenSci139.
* Active autoimmune diseases and inflammatory diseases.
* Has a history of (non-infectious) interstitial lung disease (ILD) / pneumonitis that required steroids, has current ILD / pneumonitis, or where suspected ILD / pneumonitis cannot be ruled out by imaging at screening.
* Unstable thrombotic events within 6 months prior to initiation dose of GenSci139.
* Has severe chronic or active infection
* Uncontrolled hypertension
* Has clinically significant cardiovascular disease
* Known severe hypersensitivity to GenSci139 and/or any of its excipients.
* Has a history of severe hypersensitivity reactions to other monoclonal antibodies
* With enough washout period to some therapies specified in protocol.
* Known HIV infection, active HBV or HCV infection.
* Has unresolved toxicities from previous anticancer therapy
* Had received HER2 or EGFR monoclonal antibodies, or using TOPO I inhibitor as payload, targeted to HER2 or EGFR ADC, and could not be intolerance of those treatment.
* Women who are pregnant or lactating or are planning to become pregnant.
* Uncontrollable pleural effusion, pericardial effusion, or abdominal and pelvic effusion requiring drainage and/or diuretics within 14 days prior to GenSci139 infusion.
* The other conditions of participation in this clinical trial were not considered appropriate by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2028-07-07 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part2: Incidence of adverse events | From time of informed consent to 30 days post last dose of GenSci139
  Percentage of patients with adverse events by system organ class and preferred term
Dose limiting toxicities (DLTs) | from time of first dose of GenSci139 to end of DLT observation period(approximately 21 days)
  DLTs are assessed during the DLT observation period and defined as any toxicity in DLT definition in the Clinical Study Protocol
Part1: Maximum Tolerated Dose (MTD) and Recommended Doses for Expansion (RDEs) | from time of first dose of GenSci139 up to 18 months
  To determine the maximum tolerated dose (MTD), if any, and recommend dose of expansion (RDE) for GenSci139
Part2: Objective response rate(ORR) | approximately 12 months
  To evaluate the preliminary anti-tumor activities of GenSci139 as measured by ORR using RECIST criteria v1.1.
Part2: disease control rate (DCR) | approximately 12 months
  To evaluate the preliminary anti-tumor activities of GenSci139 as measured by DCR using RECIST criteria v1.1.
Part2: Duration of response (DoR) | approximately 24 months
  To evaluate the preliminary anti-tumor activities of GenSci139 as measured by DoR using RECIST criteria 1.1.

SECONDARY OUTCOMES:
Cmax of GenSci139 | approximately 24 months
  Calculate maximum observed concentration of GenSci139
Part1: Cmax of total antibody | approximately 24 months
  Calculate maximum observed concentration of total antibody
Part1: Cmax of free payload | approximately 24 months
  Calculate maximum observed concentration of free payload
Part1: Tmax of GenSci139 | approximately 24 months
  Calculate time of maximum observed concentration of GenSci139
Part1: Tmax of total antibody | approximately 24 months
  Calculate time of maximum observed concentration of total antibody
Part1: Tmax of free payload | approximately 24 months
  Calculate time of maximum observed concentration of free payload
Part1: AUC of GenSci139 | approximately 24 months
  Calculate area under the curve of GenSci139
Part1: AUC of total antibody | approximately 24 months
  Calculate area under the curve of total antibody
Part1: AUC of free payload | approximately 24 months
  Calculate area under the curve of free payload
Part1: Objective response rate(ORR) | approximately 12 months
  To evaluate the preliminary anti-tumor activities of GenSci139 as measured by ORR using RECIST criteria v1.1.
Part1: disease control rate (DCR) | approximately 12 months
  To evaluate the preliminary anti-tumor activities of GenSci139 as measured by DCR using RECIST criteria v1.1.
Part1: Duration of response (DoR) | approximately 24 months
  To evaluate the preliminary anti-tumor activities of GenSci139 as measured by DoR using RECIST criteria 1.1.
Part1: ADA of GenSci139 | approximately 24 months
  Incidence and titer of anti-drug antibody (ADA)
Part1: NAb of GenSci139 | approximately 24 months
  Incidence and titer of neutralizing antibody (NAb)
Part2: Cmax of GenSci139 | approximately 24 months
  Calculate maximum observed concentration of GenSci139
Part2: Cmax of total antibody | approximately 24 months
  Calculate maximum observed concentration of total antibody
Part2: Cmax of free payload | approximately 24 months
  Calculate maximum observed concentration of free payload
Part2: Tmax of GenSci139 | approximately 24 months
  Calculate time of maximum observed concentration of GenSci139
Part2: Tmax of total antibody | approximately 24 months
  Calculate time of maximum observed concentration of total antibody
Part2: Tmax of free payload | approximately 24 months
  Calculate time of maximum observed concentration of free payload
Part2: AUC of GenSci139 | approximately 24 months
  Calculate area under the curve of GenSci139
Part2: AUC of total antibody | approximately 24 months
  Calculate area under the curve of total antibody
Part2: AUC of free payload | approximately 24 months
  Calculate area under the curve of free payload
Part2: ADA of GenSci139 | approximately 24 months
  Incidence and titer of anti-drug antibody (ADA)
Part2: NAb of GenSci139 | approximately 24 months
  Incidence and titer of neutralizing antibody (NAb)

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong, China